CLINICAL TRIAL: NCT00104845
Title: Injection of AJCC Stage IIB, IIC, III, and IV Melanoma Patients With Human and Mouse gp100 DNA: A Phase I Trial to Assess Safety and Immune Response
Brief Title: Vaccine Therapy in Treating Patients With Stage IIB, Stage IIC, Stage III, or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 03-007; P30CA008748 (NIH); MSKCC-IRB-03007
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

ARMS (2):
- human gp100 DNA vaccine (Experimental): Patients receive human gp100 DNA vaccine intramuscularly (IM) once in weeks 1, 4, and 7. Patients then receive mouse gp100 DNA vaccine IM once in weeks 10, 13, and 16.
  Interventions: Biological: human gp100 plasmid DNA vaccine; Biological: mouse gp100 plasmid DNA vaccine
- mouse gp100 DNA vaccine (Experimental): Patients receive mouse gp100 DNA vaccine IM once in weeks 1, 4, and 7. Patients then receive human gp100 DNA vaccine IM once in weeks 10, 13, and 16
  Interventions: Biological: human gp100 plasmid DNA vaccine; Biological: mouse gp100 plasmid DNA vaccine

INTERVENTIONS:
Biological: human gp100 plasmid DNA vaccine
Biological: mouse gp100 plasmid DNA vaccine

SUMMARY:
RATIONALE: Vaccines made from DNA may make the body build an effective immune response to kill tumor cells.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with stage IIB, stage IIC, stage III, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of vaccination with human and mouse gp100 DNA in patients with stage IIB, IIC, III, or IV melanoma.
* Determine the maximum tolerated dose of this regimen in these patients.
* Compare the antibody and T-cell response in patients treated with two different vaccination schedules.

Secondary

* Assess antitumor response in patients treated with this regimen.

OUTLINE: This is a randomized, crossover, dose-escalation study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive human gp100 DNA vaccine intramuscularly (IM) once in weeks 1, 4, and 7. Patients then receive mouse gp100 DNA vaccine IM once in weeks 10, 13, and 16.
* Arm II: Patients receive mouse gp100 DNA vaccine IM once in weeks 1, 4, and 7. Patients then receive human gp100 DNA vaccine IM once in weeks 10, 13, and 16.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 6-9 patients (at least 3 per treatment arm) receive escalating doses of human and mouse gp100 DNA vaccines until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 9 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed at 3 weeks and then annually for 15 years.

PROJECTED ACCRUAL: Approximately 18-27 patients will be accrued for this study within 6-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Stage IIB, IIC, III, or IV disease

    * Patients with stage III or IV disease who are free of disease after surgical resection* are eligible
* Patients free of disease after surgical resection* must have refused high-dose interferon alfa OR experienced recurrent disease during prior treatment with interferon alfa NOTE: *Patients who underwent surgical resection must have had the surgery within the past year
* HLA-A0201 positive
* No detectable brain metastases

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* No active bleeding

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Albumin ≥ 3.5 g/dL
* AST and ALT ≤ 2.5 times ULN
* Lactate dehydrogenase ≤ 2 times ULN
* No clinical history of hepatitis B or C

Renal

* Creatinine ≤ 2.0 mg/dL

Immunologic

* No clinical history of HIV
* No clinical history of HTLV-1
* No active infection requiring antibiotics within the past 72 hours
* No history of collagen vascular, rheumatologic, or other autoimmune disorder
* No grade 1 fever within the past 72 hours

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight ≥ 25 kg
* No serious underlying medical condition that would preclude study participation
* No preexisting uveal or choroidal eye disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 4 weeks since prior immunotherapy
* No prior immunization with any class of vaccine containing gp100, including whole cell, shed antigen, or cell lysate vaccines

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy

* No concurrent corticosteroids that would preclude study participation

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* Recovered from all prior therapy
* No other concurrent medication that would preclude study participation
* No other concurrent investigational agents
* No other concurrent systemic therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
safety and feasibility | 2 years

SECONDARY OUTCOMES:
maximum tolerated dose | 2 years
antibody and T-cell response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jedd D. Wolchok, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States